CLINICAL TRIAL: NCT00547885
Title: Randomized Controlled Double Blind Trial of Short vs Long Acting Dihydrocodeine in Chronic Non-Malignant Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPI 07-002; 2007-003639-22 (EudraCT Number)
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Pain
Keywords: dihydrocodeine; opioids, long acting; opioids, short acting; Chronic pain; non-malignant pain
MeSH Terms: conditions — Pain; Chronic Pain | interventions — dihydrocodeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Active dihydrocodeine, long acting and Placebo dihydrocodeine short acting
  Interventions: Drug: Dihydrocodeine
- 2 (Active Comparator): Placebo dihydrocodeine, long acting and active dihydrocodeine short acting.
  Interventions: Drug: Dihydrocodeine

INTERVENTIONS:
Drug: Dihydrocodeine — Group 1: 2* 60 mg dihydrocodeine long acting + up to four placebo short action
  Group 2: 3* 60 mg dihydrocodeine long acting + up to six placebo short action
  Group 3: 4* 60 mg dihydrocodeine long acting + up to eight placebo short action
  Group 4: 2 placebo for long acting + up to 4*30 mg dihydrocodeine short acting
  Group 5: 3 placebo for long acting + up to 6*30 mg dihydrocodeine short acting
  Group 6: 3 placebo for long acting + up to 8*30 mg dihydrocodeine short acting

SUMMARY:
We wish to compare the effect of long acting vs short acting opioids in chronic non-malignant pain. The study opioid is Dihydrocodeine Continus and Dihydrocodeine 30 mg tablets. We measure pain relief, health related quality of life, sleep, breakthrough pain and depression with validated questionnaires to compare the two treatment arms.

Hypothesis: The pain relief will be better and more stable with long acting opioids. Quality of sleep, breakthrough pain and quality of life will also be improved with long acting dihydrocodeine.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain
* Use 5-10 P.Forte every day for the last two weeks
* 18-75 years.

Exclusion Criteria:

* Cancer
* Hepatic failure
* Severe mental disorders
* History of known substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pain | 9 weeks
  Validated questionaires which have been properly translated to Norwegian will be used in the assessment of each outcome variable:Pain, Quality and duration of sleep, Quality of life, Depression, Moods and breakthrough pain will be measured.

SECONDARY OUTCOMES:
sleep quality and duration | 9 weeks
  Validated questionaires which have been properly translated to Norwegian will be used in the assessment of each outcome variable:Pain, Quality and duration of sleep, Quality of life, Depression, Moods and breakthrough pain will be measured.
quality of life | 9 weeks
  Validated questionaires which have been properly translated to Norwegian will be used in the assessment of each outcome variable:Pain, Quality and duration of sleep, Quality of life, Depression, Moods and breakthrough pain will be measured.
Depression and moods | 9 weeks
  Validated questionaires which have been properly translated to Norwegian will be used in the assessment of each outcome variable:Pain, Quality and duration of sleep, Quality of life, Depression, Moods and breakthrough pain will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Petter C Borchgrevink, PhD, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- National Competency Centre for Complex Disorders, Trondheim, Sør-Trøndelag, Norway

REFERENCES:
- [Result] Pedersen L, Borchgrevink PC, Breivik HP, Fredheim OMS. A randomized, double-blind, double-dummy comparison of short- and long-acting dihydrocodeine in chronic non-malignant pain. Pain. 2014 May;155(5):881-888. doi: 10.1016/j.pain.2013.12.016. Epub 2013 Dec 15. PMID 24345428